CLINICAL TRIAL: NCT03288922
Title: Comparison of Protein-bound Toxins Removals Between Limited Blood Flow Online Hemodiafiltration Using Super High-flux Dialyzer and High-Efficiency Online Hemodiafiltration With High-flux Dialyzer: An Randomized Crossover Trial
Brief Title: Protein-bound Toxin Removal Between Limited Blood Flow Super High-flux Online HDF and High-Efficiency Online HDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 291/58
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: End-stage Renal Disease; Hemodialysis
Keywords: Online Hemodiafiltration; Super high-flux dialyzer; Protein-bound uremic toxin; P-cresol
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited BF OL-HDF with SHF (Experimental): Limited blood flow pre-dilution online hemodiafiltration using super high-flux dialyzer which had larger pore size than standard high-flux dialyzer was assigned as the new intervention to compare the efficacy of protein-bound toxin removals with the control period.
  Interventions: Procedure: Limited BF OL-HDF with SHF
- High-efficiency OL-HDF (Active Comparator): High-efficiency post-dilution online hemodiafiltration using standard high-flux dialyzer was assigned as the control period.
  Interventions: Procedure: High-efficiency OL-HDF

INTERVENTIONS:
Procedure: Limited BF OL-HDF with SHF — The new modality "Limited BF OL-HDF with SHF" were performed using Fresenius 5008 hemodiafiltration machine. The prescribed blood flow rate was 300 ml/min and the total dialysis fluid flow rate was 800 ml/min which included pre-filter substitution rate of 150 ml/min. The super high-flux dialyzer was PES-17Dα from Nipro Corporation, Japan which contains 1.7 m2 hollow fiber polyethersulfone membrane (ultrafiltration coefficient 80 ml/h/mmHg; urea clearance 267 ml/min, Qb 300 ml/min and Qd 500ml/min). The patients were received this treatment thrice-a-week for 2 week before entering the wash-out period and crossover to another arm.
  Arms: Limited BF OL-HDF with SHF
Procedure: High-efficiency OL-HDF — The controlled modality "High-efficiency OL-HDF" were performed using Fresenius 5008 hemodiafiltration machine. The prescribed blood flow rate was 400 ml/min and the total dialysis fluid flow rate was 800 ml/min which included post-filter substitution rate of 100 ml/min. The standard high-flux dialyzer that was used was HF80s from Fresenius Medical Care, Germany contains 1.8 m2 hollow fiber polysulfone membrane (ultrafiltration coefficient 55 ml/h/mmHg; urea clearance 248 ml/min, Qb 300ml/min and Qd 500 ml/min). The patients were received this treatment thrice-a-week for 2 week before entering the wash-out period and crossover to another arm.
  Arms: High-efficiency OL-HDF

SUMMARY:
High-efficiency post-dilution online hemodiafiltration (OL-HDF) using high-flux dialyzer and requiring high blood flow rate (BF ≥400 mL/min) has been reported to enhance protein-bound toxin and middle molecular toxin removal and improve patient survival. Unfortunately, the majority of patients could not reach that high BF because of vascular access issue. This randomized crossover study was conducted to compare these uremic toxin removals between the new modality (limited BF OL-HDF with super high-flux dialyzer) and the control (high-efficiency OL-HDF). The OL-HDF patients were randomized to undergo either new modality or control for 2 weeks before crossover to the other modality for another 2 weeks.

DETAILED DESCRIPTION:
Elevated protein-bound toxins including p-cresol (pCS) and indoxyl sulfate (IDS) as well as middle-molecular toxins such as beta2-microglobulin (B2M) which could not be removed by hemodialysis (HD) are obviously correlated with high mortality. High-efficiency post-dilution online hemodiafiltration (OL-HDF) using high-flux dialyzer and requiring high blood flow rate (BF ≥400 mL/min) has been reported to enhance pCS, IDS, and B2M removal and improve patient survival. Unfortunately, the majority of patients could not reach that high BF because of vascular access issue. We innovated the OL-HDF modality for this limited BF situation by integrating the novel super high-flux membrane dialyzer (SHF; PES-17Dα, Nipro Corporation, Japan) into pre-dilution OL-HDF. This randomized crossover study was conducted to compare the uremic toxin removals between the new modality (limited BF OL-HDF with SHF) and the control (high-efficiency OL-HDF). The OL-HDF patients were randomized to undergo either new modality or control for 2 weeks before crossover to the other modality for another 2 weeks. Removals of pCS and IDS as well as small and middle molecule toxins were compared. The pCS and IDS were measured by high performance liquid chromatography. The dialysate albumin loss and patient safety were also monitored.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients treated with thrice-a-week OL-HDF for at least 6 months
* Residual urine < 100 mL/day

Exclusion Criteria:

* Active cardiovascular disease
* Active malignancy
* Pregnancy
* Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
pCS percentage of reduction ratio | At time 0-hour and 4-hour of the study online hemodiafiltration session
  Blood samples were taken from patients before and at the end of 4-hour in the first dialysis session of each modality. pCS levels were measured by high-performance liquid chromatography (HPLC). The percentage of reduction ratio were calculated from the before and ending samples.

SECONDARY OUTCOMES:
IDS percentage of reduction ratio | At time 0-hour and 4-hour of the study online hemodiafiltration session
  Blood samples were taken from patients before and at the end of 4-hour in the first session of each modality. IDS levels were measured by high-performance liquid chromatography (HPLC). The percentage of reduction ratio were calculated from the before and ending samples.
Beta2-microglobulin percentage of reduction ratio | At time 0-hour and 4-hour of the study online hemodiafiltration session
  Blood samples were taken from patients before and at the end of 4-hour in the first dialysis session of each modality. The percentage of reduction ratio were calculated from the before and ending samples.
Albumin loss in spent dialysate | During 4 hours of online hemodiafiltration session
  Continuous sampling of spent effluent dialysate and ultrafiltrate were carried out with a collection pump inserted into the effluent outlet line via a special connector for total albumin loss determination.

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, MD, Principal Investigator — Chulalongkorn University; Wanjak Pongsittisak, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand